CLINICAL TRIAL: NCT04919967
Title: Online Training for Addressing Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Praxis, Inc. (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nancy Byatt, Executive Director, Lifeline for Families Center & Lifeline for Moms Program;Associate Professor of Psychiatry, Obstetrics & Gynecology and Population & Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00017480; R42MH113381 (NIH)
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Mood Disorders; Anxiety Disorders
Keywords: Detection; Screening; Treatment; Depression; Anxiety; mood disorders; perinatal; maternity care
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual implementation protocol (Experimental): Participants assigned to the virtual implementation protocol plus e-learning/toolkit group will take the e-learning course an also receive support through the Virtual Implementation Protocol.
  Interventions: Behavioral: Virtual implementation protocol; Behavioral: e-learning toolkit
- E-learning/toolkit alone (Active Comparator): Participants assigned to the e-learning/toolkit alone group will only complete the e-learning course/receive the e-learning toolkit.
  Interventions: Behavioral: e-learning toolkit
- Treatment as usual (No Intervention): Participants assigned to this group will not be provided any additional training or implementation assistance. They will be able to take trainings outside of study protocol if they would otherwise plan or want to do so. They will be offered the study-specific training and implementation assistance after they have completed the final study assessments.

INTERVENTIONS:
Behavioral: Virtual implementation protocol — Participants assigned to the virtual implementation protocol plus e-learning/toolkit group will take the e-learning course and also receive additional assistance through Virtual Implementation support. The Virtual Implementation strategy will be provided through virtual assistance, training, and toolkits to help obstetric practices integrate perinatal mental health and obstetric care and is delivered over 2-3 months and includes two 1-hour virtual implementation e-meetings. Implementation will occur within the practice where a champion is identified who establishes a quality improvement team to implement the practice's change plan to achieve their goals of addressing perinatal mental health conditions.
  Arms: Virtual implementation protocol
Behavioral: e-learning toolkit — A toolkit given to obstetric care providers to enhance knowledge about and screening for perinatal mood and anxiety disorders. Participants assigned to the e-learning/toolkit alone group will take an e-learning course.This four-part online learning course aims to help obstetric care practitioners address perinatal mental health conditions such as depression, anxiety, PTSD and bipolar disorder.
  Arms: E-learning/toolkit alone; Virtual implementation protocol

SUMMARY:
The study team is developing an e-learning course to train obstetric providers to address perinatal mood and anxiety disorders. The study team will conduct a formative evaluation of the e-learning course with 10 obstetric providers and revise/refine the course based on feedback and then conduct a summative evaluation using a cluster Randomized Controlled Trial (RCT). The three-arm cluster RCT will evaluate the effectiveness of 1) a virtual implementation protocol and e-learning/toolkit as compared to 2) e-learning/toolkit alone as compared to 3) treatment-as-usual. Effectiveness will be evaluated based on rates and quality of care for perinatal mood and anxiety disorders. Using 2:2:1 randomization, the study team will randomize a minimum of 15 to a maximum of 25 obstetric practices into three groups: (1) virtual implementation protocol plus e-learning/toolkit (n=6 to 10); (2) e-learning/toolkit alone (n=6 to 10); and (3) treatment-as-usual (n=3 to 5), which will yield a maximum of 1000 patient charts evaluated for care received from obstetric providers in the randomized practices. Charts from 40 patients per practice will be evaluated at 3 different time points.

DETAILED DESCRIPTION:
The objective of this cluster RCT is to evaluate the effectiveness of adding an implementation protocol to the e-learning/toolkit in comparison to the e-learning/toolkit alone in comparison to treatment-as-usual among a maximum of 1000 patients receiving care from 15 - 25 obstetric practices regarding the rates and quality of care for perinatal mood and anxiety disorders. Using 2:2:1 randomization, we will randomize 15 - 25 obstetric practices into three groups: (1) virtual implementation protocol plus e-learning/toolkit (n=6 - 10); (2) e-learning/toolkit alone (n=6 - 10); and (3) treatment-as-usual (n=3 - 5).

The study team will conduct a baseline practice and provider assessment which will inform restricted randomization based on existing approaches to screening for perinatal mood and anxiety disorders and the clinical care of perinatal women who screen positive. Pre- and post-intervention data will be obtained through individual provider surveys to evaluate perinatal mood and anxiety disorder care practices, knowledge, and attitudes. Rates and quality of care for perinatal mood and anxiety disorders will be assessed pre- and post- using our established approach and tool to evaluate practice readiness to evaluate and address perinatal mood and anxiety disorders (Masters et al., submitted). Our tool quantifies the extent to which assessment, treatment, monitoring, and transfer of care for perinatal mood and anxiety disorders is documented in patient medical records and provides benchmarks to measure the extent to which obstetric practices successfully integrate perinatal mental health care into their workflow over time. Records will be reviewed from the initiation of prenatal care through postpartum care for given pregnancies, for all abstracted charts.

Participants in all phases of the project will complete the following: (1) a demographic questionnaire (pre-), (2) a knowledge test (pre- ,post- and final post assessment), (3) a practices and attitudes survey (pre-, post- and final post assessment), and (4) chart abstraction (pre- and post-) . The participants in the virtual implementation protocol plus e-learning/toolkit and e-learning/toolkit alone group will also complete a usability and satisfaction survey (post-test). All practices will also be asked to facilitate a medical record review/chart abstraction of a total of 120 patient files, 40 pre-pandemic and 40 post pandemic first wave and 40 post e-learning/implementation.

ELIGIBILITY:
Inclusion Criteria:

* licensed independent providers e.g. Ob/Gyn attendings and residents, family medicine, Maternal Fetal Medicine physicians (attending/fellow), certified nurse midwives, nurse practitioners, and physician assistants)

Exclusion Criteria:

* providers from the participating practices that are unable to consent,
* individuals who are not yet adults,
* prisoners
* non-English speaking participants in the study.

Pregnant women will not be excluded from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in rates of screening for bipolar disorder during the 1st or 2nd half of pregnancy. | Baseline and 13 months post baseline
  Occurrence of bipolar screening will be assessed from medical records using an established tool that evaluates practice readiness to evaluate and address perinatal mood and anxiety disorders. The extent to which screening for bipolar disorder is documented in patient medical records will be quantified. Medical records will be reviewed from the initiation of prenatal care through postpartum care for given pregnancies.

SECONDARY OUTCOMES:
Change in rates of screening for anxiety disorder during the 1st or 2nd half of pregnancy | Baseline and 13 months post baseline
  Occurrence of anxiety screening will be assessed from medical records using an established tool that evaluates practice readiness to evaluate and address perinatal mood and anxiety disorders. The extent to which screening for anxiety disorder is documented in patient medical records will be quantified. Medical records will be reviewed from the initiation of prenatal care through postpartum care for given pregnancies.
Change in Providers' quality of care for perinatal mood and anxiety disorders | Baseline and 13 months
  The documented care received by patients for perinatal mood and anxiety disorders will be measured from medical records using an established tool which rates five components in the care pathway of perinatal mood and anxiety disorders: detection, assessment, treatment initiation, follow-up & monitoring and ongoing care. Each component makes up 20% of the overall score for provider documentation/quality of care in addressing perinatal mood and anxiety disorders.

OTHER OUTCOMES:
Change in Provider Self-Reported rate of Screening | Baseline, 1 month and 13 months
  Providers are given a questionnaire to estimate their frequency of screening for perinatal mood and anxiety disorders.
Change in Provider Subject Matter Knowledge acquisition and retention | Baseline, 1 month and 13 months
  Providers are given a multiple-choice assessment to gauge provider knowledge about perinatal mood and anxiety disorders at baseline, and then provider knowledge about the subject matter post-training (at 1 month) and then retention of knowledge at 13 months.
Change in Provider attitudes and beliefs related to perinatal mood and anxiety disorders | Baseline, 1 month and 13 months
  Providers are given a questionnaire to evaluate their attitudes and believes related to perinatal mood and anxiety disorders.
Training satisfaction and usability | 1 month
  Providers are asked about their opinions of usability and satisfaction with the training course.
  Providers are asked to provide a score on a scale of their opinion, with 0 being unusable and [5] being very useable.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Byatt, DO, MS, MBA, FACLP, Principal Investigator — University of Massachusetts Medical School/UMass Memorial Health; Tiffany Moore Simas, MD, MPH, MEd, FACOG, Principal Investigator — University of Massachusetts Medical School/UMass Memorial Health
Locations (1):
- Montachusett Women's Health - UMass Memorial Health Alliance, Leominster, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is via the National Institute of Mental Health (NIMH) Data Archive (NDA) (https://ndar.nih.gov/), specifically the National Database for Clinical Trials Related to Mental Illness (NDCT).
Time Frame: Data will be deposited into the NDCT repository as soon as possible but no later than within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier. We will adhere to the NIH Data Sharing Policy and Implementation Guidance.
Access Criteria: The data will be deposited and made available through NDCT, which is an NIH-funded repository, and that these data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary studies related to perinatal mental health.
  Final research data and data communication will be available to researchers under an appropriate data sharing agreement that provides for: (1) use of data only for research purposes (and not to identify any individual participant); (2) securing the data using appropriate measures; (3) not redistributing the data; (4) destroying or returning the data after analyses are completed; (5) not using the data for commercial purposes; and (6) proper acknowledgement of the data source.
  All data products can be transferred to approved investigators by secure encrypted transfer using the secure managed data transfer server, MoveIt DMZ (Ipswitch File Transfer Inc.).

REFERENCES:
- [Background] McLaughlin TJ, Aupont O, Kozinetz CA, Hubble D, Moore-Simas TA, Davis D, Park C, Brenner R, Sepavich D, Felice M, Caviness C, Downs T, Selwyn BJ, Forman MR. Multilevel Provider-Based Sampling for Recruitment of Pregnant Women and Mother-Newborn Dyads. Pediatrics. 2016 Jun;137 Suppl 4(Suppl 4):S248-57. doi: 10.1542/peds.2015-4410F. PMID 27251871
- [Background] Johnson JE, Wiltsey-Stirman S, Sikorskii A, Miller T, King A, Blume JL, Pham X, Moore Simas TA, Poleshuck E, Weinberg R, Zlotnick C. Protocol for the ROSE sustainment (ROSES) study, a sequential multiple assignment randomized trial to determine the minimum necessary intervention to maintain a postpartum depression prevention program in prenatal clinics serving low-income women. Implement Sci. 2018 Aug 22;13(1):115. doi: 10.1186/s13012-018-0807-9. PMID 30134941
- [Background] Byatt N, Moore Simas TA, Biebel K, Sankaran P, Pbert L, Weinreb L, Ziedonis D, Allison J. PRogram In Support of Moms (PRISM): a pilot group randomized controlled trial of two approaches to improving depression among perinatal women. J Psychosom Obstet Gynaecol. 2018 Dec;39(4):297-306. doi: 10.1080/0167482X.2017.1383380. Epub 2017 Oct 10. PMID 28994626
- [Background] Byatt N, Pbert L, Hosein S, Swartz HA, Weinreb L, Allison J, Ziedonis D. PRogram In Support of Moms (PRISM): Development and Beta Testing. Psychiatr Serv. 2016 Aug 1;67(8):824-6. doi: 10.1176/appi.ps.201600049. Epub 2016 Apr 15. PMID 27079994
- [Background] Ivers NM, Halperin IJ, Barnsley J, Grimshaw JM, Shah BR, Tu K, Upshur R, Zwarenstein M. Allocation techniques for balance at baseline in cluster randomized trials: a methodological review. Trials. 2012 Aug 1;13:120. doi: 10.1186/1745-6215-13-120. PMID 22853820
- [Background] Tajima B, Guydish J, Delucchi K, Passalacqua E, Chan M, Moore M. Staff Knowledge, Attitudes, and Practices Regarding Nicotine Dependence Differ by Setting. J Drug Issues. 2009;39(2):365-384. doi: 10.1177/002204260903900208. PMID 20617124
- [Background] Moore Simas TA, Brenckle L, Sankaran P, Masters GA, Person S, Weinreb L, Ko JY, Robbins CL, Allison J, Byatt N. The PRogram In Support of Moms (PRISM): study protocol for a cluster randomized controlled trial of two active interventions addressing perinatal depression in obstetric settings. BMC Pregnancy Childbirth. 2019 Jul 22;19(1):256. doi: 10.1186/s12884-019-2387-3. PMID 31331292